CLINICAL TRIAL: NCT06572007
Title: Relationships of Fascia Thickness With Pain, Flexibility, Disability and Depression in Individuals With Chronic Low Back Pain
Brief Title: The Impact Of Fascia Thickness on Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Emine Atıcı, Principal Investigator, Okan University
Other Study IDs: 26.10.2022/159
Record Dates: First submitted 2024-08-20; First posted 2024-08-26 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain; Disability Physical; Pain, Chronic
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Low back pain: Fascia thickness of individuals with chronic low back pain will be measured by ultrasound and the relationship with pain, flexibility, disability and depression will be analysed.
  Interventions: Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Ultrasound — To investigate the thickness of the fascia tissue, the subjects will undergo an ultrasound examination using a clinical ultrasound system (S9, SonoScape Corporation, made in China) with a linear 5-14 MHz array of L14-5/38. The transducer with a cross-section of 6.24 cm2 will be aimed at points 2 cm lateral to the midline of the L2 and L3 vertebrae on both sides of the spine.

SUMMARY:
This study aimed to investigate the impact of lumbar perimuscular and subcutaneous zone thickness on pain, functionality, disability, and depression in individuals with chronic low back pain (CLBP).

DETAILED DESCRIPTION:
This study investigates the role of the thoracolumbar fascia (TLF) in chronic low back pain (CLBP) persisting for more than one year. Specifically, the researchers aim to examine the relationships between various factors in individuals with CLBP, including the thickness of the perimuscular and subcutaneous regions in the lumbar and hamstring regions. The relationship with functional tests of the lower back and lower limbs will also be analysed. In addition, the intensity of the pain experienced by the participants, the extent to which the pain restricts their daily activities, and depression scores will be assessed. Through this analysis, the researchers aim to gain a deeper understanding of TLF's involvement in CLBP and its impact on the overall well-being of affected individuals.

ELIGIBILITY:
Inclusion Criteria:

* The absence of LBP in the last 12 months,
* A body mass index (BMI) of 18.5 to 30,
* An age between 30 and 50 years.

Exclusion Criteria:

* History of musculoskeletal diseases,
* a history of back and lower limb surgery,
* the use of anti-inflammatory drugs and steroids

Ages: 30 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Getting a diagnosis of low back pain
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | baseline
  The Visual Analog Scale, a 100 mm long scale marked at every 10 mm and ranging from 0 to 10, will be used to assess the level of pain. Patients mark their own pain level on this scale, scoring between 0 and 10, where 0 indicates "no pain" and 10 represents "the worst possible pain"
Straight Leg Raise Test (SLR) | baseline
  The Straight Leg Raise Test is a physiotherapy method used to determine the range of motion of the hip joint. The patient lies supine. They are instructed to lift one leg as high as possible without bending the knee. The leg that remains on the ground should not lift, and its knee should remain extended. The point reached by the raised leg is measured with a goniometer. The same procedure is repeated for the other leg . Normally, the hip flexion angle is 90 degrees; a range of 70-90 degrees is considered normal in adults. An angle below 70 degrees indicates restriction.
Lumbar Extensor Shortening Assessment | baseline
  This physiotherapy method is used to evaluate the shortening of the extensor muscles in the lumbar region. The patient lies supine with their arms in a reverse 'T' position. They are instructed to flex both hips and knees and draw them towards their abdomen. The distance between the knees and the chest is recorded

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire (RMDQ) | baseline
  The Turkish version of the Roland Morris Disability Questionnaire will be used to measure disability. The RMDQ, first published in 1983, assesses the disability level of individuals with back pain(23). It consists of 24 items, including physical ability/activity (15 items), sleep/rest (3 items), psychosocial (2 items), home management (2 items), eating (1 item), and pain frequency (1 item). The original 24-item questionnaire has been shortened to 18-item and 23-item versions and adapted for use in other countries . It was adapted into Turkish by Küçükdeveci et al. in 2001. Each positive response corresponds to one point on the scale, addressing daily activities potentially restricted by back pain. Each "Yes" answer scores 1 point, and each "No" answer scores 0 points, with the final score being the sum of these points. The total score ranges from 0 to 24, with higher scores indicating greater disability .
Beck Depression Inventory | baseline
  The Turkish version of the Beck Depression Inventory, developed by Beck and colleagues, will be used. Adapted into Turkish by Hisli N. in 1988, the inventory consists of 21 questions, each separately scored to obtain a total score. The possible scores range from 0 to 63. Scores of 0-9 indicate minimal depression, 10-16 mild depression, 17-29 moderate depression, and 30-63 severe depression

CONTACTS AND LOCATIONS:
Overall Officials: Emine Atıcı, Study Director — Okan University
Locations (2):
- Turkey (Türkiye) (2):
  - Emine Atıcı, Tuzla, Istanbul
  - Istanbul Okan University, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided